CLINICAL TRIAL: NCT01707433
Title: Diagnosis of Mucopolysaccharidosis Disorders in Patients Presenting With Bilateral Hip Disease
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: BioMarin Pharmaceutical (Industry); Greenwood Genetic Center (Other); Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Nancy Mendelsohn, Medical Director of Genetic Dept, Children's Hospitals and Clinics of Minnesota
Other Study IDs: MPSHIP
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Mucopolysaccharidosis IV A; Mucopolysaccharidosis VI
Keywords: spondyloepiphyseal dysplasia; multiple epiphyseal dysplasia; bilateral Legg Calve Perthes; bilateral proximal femoral epiphyseal dysplasia; GALNS
MeSH Terms: conditions — Mucopolysaccharidosis IV; Mucopolysaccharidosis VI; Osteochondrodysplasias | interventions — Clinical Enzyme Tests

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnosis of hip disease: Diagnosed with spondyloepiphyseal dysplasia or multiple epiphyseal dysplasia or bilateral Legg-Calve-Perthes disease, or bilateral proximal femoral epiphyseal dysplasia
  Interventions: Other: Enzyme testing

INTERVENTIONS:
Other: Enzyme testing — Leukocyte activity measurement of Arylsulfatase B and N acetyl galactosamine 6 sulfatase (GALNS)

SUMMARY:
BACKGROUND/OBJECTIVE: Quantitative urine screening for mucopolysaccharides (MPS) has been the primary method for detecting mucopolysaccharidoses in children. This method may not be sufficiently sensitive and may miss some patients with arylsulfatase B (ARSB) deficiency. Investigators propose to identify patients retrospectively and prospectively who carry a diagnosis of spondyloepiphyseal dysplasia, multiple epiphyseal dysplasia, bilateral proximal femoral epiphyseal dysplasia, or bilateral Legg-Calve-Perthes. For these patients, investigators will perform enzyme testing on a blood sample which will identify MPS VI or IVA.

Patients who have an earlier diagnosis of MPS are likely to have better health outcomes with medical management. Therefore, it is important to determine effective diagnostic methods. Investigators believe that bilateral hip involvement should alert the clinician to the possibility of MPS VI and further examination. The purpose of this study is to test the hypothesis that the correct diagnoses of two MPS storage disorders are delayed in patients with bilateral proximal femoral epiphyseal dysplasia and normal quantitative urine MPS studies.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 21 years of age
* Diagnosis of spondyloepiphyseal dysplasia or multiple epiphyseal dysplasia or bilateral Legg-Calve-Perthes disease or bilateral proximal femoral epiphyseal dysplasia.

Exclusion Criteria:

* Definitive etiology for above-mentioned diagnosis (i.e. other MPS disease, known chondrodysplasia, Meyer's dysplasia)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Males/females less than or equal to 21 years of age who have been seen at Gillette Children's Specialty Healthcare or Children's Hospitals and Clinics of Minnesota and carry a diagnosis of spondyloepiphyseal dysplasia or multiple epiphyseal dysplasia or bilateral Legg-Calve-Perthes disease or bilateral proximal femoral epiphyseal dysplasia.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Subjects identified with MPS IVA or VI | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mendelsohn, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (2):
- United States (2):
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota